CLINICAL TRIAL: NCT00927524
Title: An Open-Label, Randomized, Two-Period, Crossover Study to Characterize the Insulin Exposure and Glucose Response to Meals in Type 1 Diabetic Subjects Administered Two Different Insulin Regimens Compared to the Endogenous Insulin Exposure and Glucose Response to Meals In Healthy Adult Controls
Brief Title: Insulin Exposure and Glucose Response to Meals in Type 1 Diabetic Subjects Administered Two Different Insulin Regimens Compared to the Endogenous Insulin Exposure and Glucose Response to Meals In Healthy Adult Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Steve Davis, Department Chair, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 050116
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
Keywords: Insulin analogs; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — insulin glulisine; Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apidra (insulin glulisine) (Active Comparator): Administration of Apidra at three meals during a 24 hour period.
  Interventions: Drug: Insulin glulisine
- 70/30 insulin (Active Comparator): Administration of 73/30 insulin at three meals during a 24 hour period.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin glulisine — Dose injection of insulin glargine (Lantus®) given subcutaneously in the abdomen 1 hour prior to breakfast and a dose of insulin glulisine (Apidra®) at a dose based upon your (body wt.) carbohydrate intake for each of the three meals (breakfast, lunch and dinner).
  Other Names: Apidra
  Arms: Apidra (insulin glulisine)
Drug: Insulin — Dose based on carbohydrate intake given subcutaneously in the abdomen prior to breakfast and dinner.
  Other Names: Humalog 70/30
  Arms: 70/30 insulin

SUMMARY:
Intensive control of Type 1 Diabetes is critical in prevention of long term complications. Unfortunately, there is a three-fold increase in hypoglycemia with intensive control. Hypoglycemia is often the major limiting factor in achieving good control. Insulin treatment of diabetes is composed of some form of short acting insulin regimen in order to provide control of blood glucose excursions that are the result of glucose intake as well as a basal insulin regimen either in a continuous administration (as in continuous subcutaneous insulin infusion-"pump therapy"), once a day injection (insulin Glargine), twice a day (ultralente or NPH or lente insulin) or a premixed version that is combined with the short acting insulin (70/30 or 75/25). Often low blood sugars are the result of less physiologically absorbed insulins whose peak of action is earlier or later than the peak absorption of glucose from a meal.

Apidra (glulisine insulin) is a new short acting insulin analogue whose peak and duration of action are ideal in that it may be administered more appropriately prior to and even after a meal with evidence of good control of blood glucose excursions from a meal. The purpose of this study is to compare the effect of Apidra upon meal related blood glucose profile as compared to those treated with 70/30 insulin in patients with Type 1 Diabetes. The investigators also will study healthy volunteers as controls who will not be treated with insulin but will be evaluated for mealtime absorption and blood glucose profile during similar meal intake. The investigators will use a stable isotope tritiated glucose.

DETAILED DESCRIPTION:
Intensive control of Type 1 Diabetes is critical in prevention of long term complications. Unfortunately, there is a three-fold increase in hypoglycemia with intensive control. Hypoglycemia is often the major limiting factor in achieving good control. Insulin treatment of diabetes is composed of some form of short acting insulin regimen in order to provide control of blood glucose excursions that are the result of glucose intake as well as a basal insulin regimen either in a continuous administration (as in continuous subcutaneous insulin infusion-"pump therapy"), once a day injection (insulin Glargine), twice a day (ultralente or NPH or lente insulin) or a premixed version that is combined with the short acting insulin (70/30 or 75/25). Often low blood sugars are the result of less physiologically absorbed insulins whose peak of action is earlier or later than the peak absorption of glucose from a meal.

Apidra (glulisine insulin) is a new short acting insulin analogue whose peak and duration of action are ideal in that it may be administered more appropriately prior to and even after a meal with evidence of good control of blood glucose excursions from a meal. The purpose of this study is to compare the effect of Apidra upon meal related blood glucose profile as compared to those treated with 70/30 insulin in patients with Type 1 Diabetes. We also will study healthy volunteers as controls who will not be treated with insulin but will be evaluated for mealtime absorption and blood glucose profile during similar meal intake. We will use a stable isotope tritiated glucose.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Subjects

  1. 12 adults (males or females) with Type 1 Diabetes, aged 18 to 55 years.
  2. C-peptide-negative
  3. Body mass index < 29.0 kg/m2
* Healthy Subjects

  1. 12 non-smoking adults (males or females), aged 18 to 55 years
  2. Normal response to an oral glucose tolerance test (OGTT)
  3. Body mass index < 29.0 kg/m2

Exclusion Criteria:

* Diabetic Subjects

  1. Hemoglobin A1c >9%
  2. Total daily insulin requirements >0.8 units/kg actual body weight
  3. History of hypoglycemia that required the subject to see medical attention (i.e., doctor's office visit, ER visit, or EMT/paramedic attention) within 6 months of the study.
  4. History of acute metabolic complications within 3 months of the study
  5. History of lipodystrophy.
  6. History of or suspected diabetic gastroparesis or current treatment with any drugs known to affect gastrointestinal motility.
  7. Inability or unwillingness to administer subcutaneous insulin injections in the abdomen.
  8. Any past or present clinically relevant abnormality, medical condition, or circumstance making the subject unsuitable for participation in the study.
  9. Active peptic ulcer disease or a history of gastrointestinal surgery within the last 6 months years.
  10. History of malignancy (except basal cell carcinoma and carcinoma in situ) within the last 5 years.
  11. Pregnant or lactating females or females of childbearing potential who are unwilling to abstain from sexual intercourse or use reliable, medically accepted methods of contraception.
  12. History of alcoholism or drug abuse within 12 months of the study.
  13. Is the investigator, sub-investigator, research assistant, pharmacist, study coordinator, other study staff, or relative thereof directly involved in the conduct of this protocol.
* Healthy Subjects

  1. Hemoglobin A1c >6.0%
  2. Any past or present clinically relevant abnormality, medical condition, or circumstance making the subject unsuitable for participation in the study.
  3. Historical, clinical, or laboratory evidence of liver disease including but not limited to transaminase activity concentrations >2.5 times the upper limit of the reference range.
  4. Current treatment with any drugs known to affect gastrointestinal motility.
  5. Active peptic ulcer disease or a history of gastrointestinal surgery within the last 6 months.
  6. History of malignancy (except basal cell carcinoma and carcinoma in situ) within the last 5 years.
  7. Pregnant or lactating females or females of childbearing potential who are unwilling to abstain from sexual intercourse or use reliable, medically accepted methods of contraception.
  8. History of alcoholism or drug abuse within 12 months of the study.
  9. Is the investigator, sub-investigator, research assistant, pharmacist, study coordinator, other study staff, or relative thereof directly involved in the conduct of this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2006-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Insulin levels | 24 hours